CLINICAL TRIAL: NCT06590298
Title: Evaluating the Effects of Adjunctive Aripiprazole on Weight and Metabolic Outcomes in Females Receiving Atypical Antipsychotics: a Randomized Clinical Trial
Brief Title: Evaluating the Effects of Adjunctive Aripiprazole on Weight and Metabolic Outcomes in Females
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Arshed Muhammad, PhD studentship, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UIAT
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Psychosis; Metabolic Syndrome; Weight Gain
MeSH Terms: conditions — Psychotic Disorders; Metabolic Syndrome; Weight Gain

STUDY DESIGN:
Intervention Model Description: Two-arm randomized control trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The intervention group will be added 5 mg of aripiprazole as an adjunct with the usual antipsychotic treatment to the females on antipsychotic treatment
  Interventions: Drug: Adjunctive Aripiprazole for improving Weight and Metabolic Outcomes in Females
- Control (No Intervention): No intervention will be given except usual antipsychotic treatment

INTERVENTIONS:
Drug: Adjunctive Aripiprazole for improving Weight and Metabolic Outcomes in Females — The intervention group will be added 5 mg of aripiprazole as an adjunct with the usual antipsychotic treatment to the females on antipsychotic treatment
  Arms: Intervention group

SUMMARY:
Patients with psychiatric disorders, including depression, anxiety, and schizophrenia, often require antipsychotic medications for symptom management. However, metabolic changes, especially weight gain, are a common and challenging side effect of many antipsychotics. Aripiprazole, an atypical antipsychotic, has shown promise in mitigating this adverse effect when used in combination with other antipsychotic medications.

DETAILED DESCRIPTION:
This study aims to investigate the effectiveness of different combinations of aripiprazole with atypical antipsychotics in preventing or minimizing weight gain in patients with various psychiatric conditions. While weight gain affects both genders, females may be particularly vulnerable due to physiological differences and societal pressures related to body image.

Collectively, while individual studies have specific nuances, the general trend suggests that combining Aripiprazole with dietary modifications and potentially lifestyle changes shows promise in managing weight gain associated with antipsychotic medications in females.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18-65 years diagnosed with a mental health condition necessitating antipsychotic treatment.
* Diagnosis of Schizophrenia or Schizoaffective Disorder
* On stable doses of atypical antipsychotics, either Olanzapine, Clozapine, or Risperidone for at least 1 month
* Willingness to comply with the study protocol.

Exclusion Criteria:

* Pregnancy or lactation.
* Severe medical conditions impacting weight or metabolism.
* Previous intolerance or contraindications to Aripiprazole.
* Non-compliant with prescribed medications
* Mental Retardation
* Participant with an eating disorder
* Participants with serious suicidal thoughts, or who pose a serious risk of harm to self or to others.
* Diagnosis of Hyper or Hypothyroidism; Evidence of thyroid dysfunction as evidenced by serum thyroid function tests (i.e Thyroid Stimulating Hormone and -Free Thyroxine (fT4) levels > 10 % above or below the limits of the normal range Use of any medication for weight loss within the past one month to the study entry
* Clinically significant abnormalities in physical examinations, ECG or lab assessments

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females on antipsychotic medication
Enrollment: 600 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-04-10 (Estimated)

PRIMARY OUTCOMES:
Mean change in body weight in kilograms | 6-months from baseline
  Mean change in body weight measured by digital weight machine

SECONDARY OUTCOMES:
Body Mass Index (BMI) | 6-months from baseline
  Body Mass Index (BMI) will be calculated by Body Mass Index (BMI) calculator
Metabolic markers (fasting blood glucose; HbA1c; triglycerides; total, HDL and LDL cholesterol levels) | 12 months from baseline
  Biochemical laboratory test
Change in waist circumference in cm | 6-months from baseline
  Change in waist circumference will be measured by an inch tape

CONTACTS AND LOCATIONS:
Overall Officials: MUHAMMAD ARSHED, PhD, Principal Investigator — University of Lahore

REFERENCES:
- [Background] Wang M, Tong JH, Zhu G, Liang GM, Yan HF, Wang XZ. Metformin for treatment of antipsychotic-induced weight gain: a randomized, placebo-controlled study. Schizophr Res. 2012 Jun;138(1):54-7. doi: 10.1016/j.schres.2012.02.021. Epub 2012 Mar 5. PMID 22398127
- [Background] Weiden PJ. Switching antipsychotics as a treatment strategy for antipsychotic-induced weight gain and dyslipidemia. J Clin Psychiatry. 2007;68 Suppl 4:34-9. PMID 17539698
- [Background] Cooper SJ, Reynolds GP; With expert co-authors (in alphabetical order):; Barnes T, England E, Haddad PM, Heald A, Holt R, Lingford-Hughes A, Osborn D, McGowan O, Patel MX, Paton C, Reid P, Shiers D, Smith J. BAP guidelines on the management of weight gain, metabolic disturbances and cardiovascular risk associated with psychosis and antipsychotic drug treatment. J Psychopharmacol. 2016 Aug;30(8):717-48. doi: 10.1177/0269881116645254. Epub 2016 May 4. PMID 27147592
- [Background] Carli M, Kolachalam S, Longoni B, Pintaudi A, Baldini M, Aringhieri S, Fasciani I, Annibale P, Maggio R, Scarselli M. Atypical Antipsychotics and Metabolic Syndrome: From Molecular Mechanisms to Clinical Differences. Pharmaceuticals (Basel). 2021 Mar 8;14(3):238. doi: 10.3390/ph14030238. PMID 33800403